CLINICAL TRIAL: NCT04874350
Title: A Phase 2, Randomized Double-Blind, Placebo-Controlled, Multi-Center Study to Assess the Efficacy, Safety, and Tolerability of Oral LPCN 1148 in Male Subjects With Cirrhosis of the Liver and Sarcopenia
Brief Title: A Study to Assess the Efficacy, Safety, and Tolerability of Oral LPCN 1148 in Male Subjects With Cirrhosis of the Liver and Sarcopenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lipocine Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LPCN 1148-21-001
Record Dates: First submitted 2021-05-03; First posted 2021-05-05 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Liver Cirrhosis; Sarcopenia
MeSH Terms: conditions — Liver Cirrhosis; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 to LPCN 1148 or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LPCN 1148 (Experimental): Oral LPCN 1148 capsules, administered as BID.
  Interventions: Drug: LPCN 1148
- Placebo (Placebo Comparator): Oral matching placebo capsules, administered as BID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LPCN 1148 — LPCN 1148 is an oral capsule product containing an ester prodrug of bioidentical testosterone, designed to enable absorption via intestinal lymphatics.
  Arms: LPCN 1148
Drug: Placebo — Oral matching placebo capsule
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to assess the efficacy, safety, and tolerability of LPCN 1148 in men with cirrhosis of the liver and sarcopenia.

DETAILED DESCRIPTION:
This is a 52-week, multicenter, double-blind, placebo-controlled, two arm study of LPCN 1148 in adult men with cirrhosis of the liver and sarcopenia on the liver transplant waitlist. This study will evaluate the efficacy, safety, and tolerability of LPCN 1148, determined through a range of clinical outcomes and functional and laboratory tests.

Approximately 48 subjects will be randomized 1:1 ratio to receive one of the following treatments:

* Treatment A: Oral LPCN 1148
* Treatment B: Oral matching placebo.

Subjects will undergo a screening period to determine study eligibility. Adult male subjects with liver cirrhosis and sarcopenia on the transplant list will be enrolled into the study.

There are two treatment phases to this study.

* Stage 1: 24 weeks of blinded study treatment (LPCN 1148 or matching placebo)
* Stage 2: 28-week open-label extension. Subjects who participate in Stage 1 of this trial will roll over to a 28-week open-label extension phase. All subjects will receive LPCN 1148; there will be no placebo in the extension period.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥ 18 years old
2. Currently listed, on the liver transplant waitlist for cirrhosis secondary to Hepatitis B or C infection, Alcoholic Liver Disease (ALD), Non-Alcoholic Steatohepatitis (NASH), Primary Biliary Cholangitis (PBC), or Primary Sclerosing Cholangitis (PSC)
3. Evidence of sarcopenia with appropriate cutoff recommended by clinical guidance

Exclusion Criteria:

1. Suspected or proven hepatocellular carcinoma (HCC)
2. History of current or suspected prostate or breast cancer
3. History of malignancies other than prostate, breast, or HCC, unless successfully treated with curative intent and believed to be cured (defined as complete remission lasting at least 5 years)
4. History of uncontrolled or recurrent portal hypertensive bleeding, including uncontrolled or recurrent bleeding from varices, gastropathy, colopathy, or hemorrhoidal bleeding in the past 6 months.
5. History or current thrombosis (including portal vein thrombosis), thromboembolism, or treatment for portal vein thrombosis
6. History of hemochromatosis
7. History of hypercoagulable state (e.g. Factor V Leiden deficiency, protein C deficiency, protein S deficiency, anti-thrombin III deficiency, or the presence of lupus anticoagulant)
8. Prior history of complications of ascites in the past 6 months including:

   1. Spontaneous bacterial peritonitis
   2. Hepatic hydrothorax
9. MELD score > 25
10. Abnormal lab value in serum chemistry, hematology, or urinalysis that the PI considers clinically significant, including but not limited to:

    1. PSA > 4 ng/mL
    2. Polycythemia (Hematocrit > ULN) or history of polycythemia
    3. ALT or AST > 5x ULN
    4. ALP > 2x ULN; subjects with PBC or PSC are excluded if ALP is > 10x ULN
    5. Platelet count < 30,000/mL
    6. EGFR < 30 mL/min/1.73 m2 for subjects not undergoing routine, scheduled dialysis
    7. Serum albumin < 2.0 g/dL
    8. INR > 2.3
11. Subjects with PSA between 2.5 ng/mL and 4 ng/mL are excluded only if any of the below criteria are met at baseline:

    1. Hematocrit > 48%
    2. I-PSS > 19
    3. Any irregularity found on digital rectal examination of the prostate
12. Subjects with PSA > 3 ng/mL are excluded only if any of the below criteria are met at baseline:

    1. Subject is African American
    2. Subject has a first-degree relative who has a history of prostate cancer
    3. Hematocrit > 48%
    4. I-PSS > 19
    5. Any irregularity found on digital rectal examination of the prostate
13. Clinically significant abnormal prostate digital rectal examination (DRE) in the opinion of the PI, with DRE screening initiated at International Prostate Symptom Score (I-PSS) > 19
14. History of bariatric surgery
15. History of stroke or myocardial infarction within the past 5 years
16. History of TIPS within the past 6 months, or TIPS procedure expected within 6 months of Day 1
17. Known positivity for Human Immunodeficiency Virus (HIV) infection
18. Acute liver failure as the indication for addition to the liver transplant waitlist
19. Estimated life expectancy less than 3 months or expected to undergo liver transplant within 3 months
20. Known heart failure of New York Heart Association class III or IV
21. Evidence of severe encephalopathy at screening encephalopathy that is not controlled despite adequate medical therapy
22. History of prior organ transplant
23. History of Fontan physiology
24. History of pulmonary embolus
25. Porto-pulmonary hypertension
26. Hepatopulmonary syndrome requiring standing home supplemental oxygen therapy, or MELD exception points for hepatopulmonary syndrome
27. Uncontrolled epilepsy or migraine
28. Active substance abuse or dependency extending to within the previous 3 months
29. History of significant sensitivity or allergy to testosterone, or product excipients.
30. Use of known strong inhibitors (e.g., ketoconazole) or inducers (e.g., dexamethasone, phenytoin, rifampin, carbamazepine) of cytochrome P450 3A (CYP3A) within 30 days prior to study drug administration and through the end of the study
31. Subjects who are currently receiving any androgens (testosterone or other androgens or androgen-containing supplements) and are unwilling to washout prior to screening

    a. Washout: 12 weeks following long-acting intramuscular androgen injections; 4 weeks following topical or buccal androgens; 3 weeks following oral androgens
32. Uncontrolled hypertension (>160/90 mmHg despite treatment)
33. Uncontrolled obstructive sleep apnea
34. Use of any investigational drug within 5 half-lives of the last dose or in the past 6 months prior to Study Day -2 without medical monitor and/or Sponsor approval
35. Subject who is not willing to use adequate contraception for the duration of the study
36. Any other condition, which in the opinion of the investigator would impede compliance to the study protocol (including diet, exercise, and alcohol abstinence) or hinder completion of the study
37. Failure to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Skeletal Muscle Index in LPCN 1148 treated subjects compared to placebo | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in Liver Frailty Index in LPCN 1148 treated subjects compared to placebo | 24 weeks
Change in number of breakthrough hepatic encephalopathy events in LPCN 1148 treated subjects compared to placebo | 24 weeks
  Breakthrough hepatic encephalopathy was defined as events of hepatic encephalopathy with a Common Terminology Criteria for Adverse Events grade greater than grade 1

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Mayo Clinic, Scottsdale, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Maryland Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Methodist Health System, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Mt.Olympus Medical Research, Houston, Texas
  - Intermountain Healthcare, Murray, Utah
  - University of Utah, Salt Lake City, Utah